CLINICAL TRIAL: NCT06216054
Title: A Randomized, Double-blind, Placebo-controlled, Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetic of Multiple-ascending Doses of LPM3770164 Sustained-release Tablets in Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetic of Multiple-ascending Doses of LPM3770164 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY03015/CT-CHN-102
Record Dates: First submitted 2023-12-19; First posted 2024-01-22 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Tardive Dyskinesia; Huntington Disease
MeSH Terms: conditions — Tardive Dyskinesia; Huntington Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LPM3770164 (Experimental): LPM3770164 sustained-release tablets will be administrated with multiple doses from 5mg to 30mg on day 1~10
  Interventions: Drug: LPM3770164 sustained release tablet
- Placebo (Placebo Comparator): LPM3770164 sustained release tablet simulant will be administrated on day 1~10
  Interventions: Drug: LPM3770164 sustained release tablet simulant

INTERVENTIONS:
Drug: LPM3770164 sustained release tablet — administrated orally
  Arms: LPM3770164
Drug: LPM3770164 sustained release tablet simulant — administrated orally
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, multiple-ascending doses trial to evaluate the safety, tolerability and pharmacokinetic of LPM3770164 sustained-release tablets orally administered in healthy subjects under fasting state, providing the rationale information for later clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who voluntarily participate and sign the informed consent form;
2. Healthy male/female volunteers aged 18 to 45 years;
3. Body weight ≥ 50.0 kg for men and ≥ 45.0 kg for women, and body mass index (BMI) 18.5 ~ 26.0 kg/m2, inclusive;
4. Able to comply with the lifestyle restrictions.

Exclusion Criteria:

1. Subject has a history of allergy to any component of the investigational drug or similar drugs, or allergic constitution;
2. Subject has a current or past medical history that may affect the clinical trial or dysfunction, including but not limited to the past or current respiratory system, circulatory system, digestive system, urinary system, reproductive system, nervous system, endocrine system, immune system, motor system, blood system, psychiatry/ psychology, dermatology and other clinically serious diseases or chronic diseases; or any other diseases that may interfere with the test results;
3. Any surgical condition or condition may significantly affect the absorption, distribution, metabolism and excretion of the drug, or may pose a hazard to the subjects;.
4. Subject has a history of self-mutilation; or at risk of suicide;
5. Subject has a history of surgery within 3 months prior to administration, or failure to recover from surgery, or having an expected surgical plan during the trial;
6. Subject has abnormal vital signs, laboratory abnormalities, and ECGs;
7. Subject has used any of over-the-counter products within 7 days or prescription medications within 28 days prior to dosing;
8. Subject positive for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), HIV antibody (HIV-Ab), or syphilis seroreactivity (Trust);
9. Subject has a history of alcohol abuse within 1 year or positive alcohol breath test results;
10. Subject has a history of substance abuse within 1 year or a positive urine drug screen;
11. Subject who has daily smoking of ≥ 5 cigarettes within 3 months;
12. Subject who has special requirements for food, cannot comply with the unified diet or have dysphagia;
13. Subject who has consumption of xanthine-rich foods or beverages (such as tea, coffee, cola, or chocolate) within 3 days prior to administration;
14. Subject who has consumption of food or beverages containing grapefruit within 7 days prior to administration;
15. Subject who has participated in other clinical trials within 3 months before administration;
16. Subject has used blood products or being blood donor or blood loss within 3 months;
17. Pregnant, lactating women, or positive pregnancy test;
18. Subject who refusal to contraception, or plan to donate sperm or ovums;
19. Other conditions which would make participation in the study unsuitable.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse event | from baseline to day 37
  Number of participants with treatment-emergent adverse event will be summarized by Group, System Organ Classification (SOC), Preferred Term (PT), severity and the relationship with treatment.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | from day 1 to day 24
Area Under the Curve from time 0 to 24 hours (AUC0-24) | from day 1 to day 24
Area Under the Curve from time 0 to the last measurable concentration (AUC0-t) | from day 1 to day 24
Area Under the Curve from time 0 extrapolated to infinity (AUC0-inf) | from day 1 to day 24
Time to maximum concentration (Tmax) | from day 1 to day 24
Half-life (t1/2) | from day 1 to day 24
ECG QTc Interval | from baseline to day 37

CONTACTS AND LOCATIONS:
Overall Officials: Huafang Li, Doctor, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China